CLINICAL TRIAL: NCT03347149
Title: Nurses' Customization of Physiologic Monitor Alarms: Outcomes and User Acceptance of the IntelliVue Alarm Advisor Software
Brief Title: Outcomes and User Acceptance of the IntelliVue Alarm Advisor Software (USA)
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: PMS-BBN-US-AA-2.01
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Clinical Alarms
Keywords: Alarms; Alarm Fatigue; Alarm Nuisance; Alarm Reduction; Patient Monitoring; Intensive Care
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Pre-Phase (Control): no Alarm Advisor Software installed
- Post-Phase (Observation): Alarm Advisor Software implemented
  Interventions: Device: Alarm Advisor Software

INTERVENTIONS:
Device: Alarm Advisor Software — Providing advice on alarm limits as part of routine medical care
  Groups: Post-Phase (Observation)

SUMMARY:
This Clinical Study will be conducted as a comparative study focusing on usability and efficiency by comparing alarm burden pre- and post- implementation of an "Alarm Advisor software".

DETAILED DESCRIPTION:
In a first phase of data collection (pre-implementation) all alarms of an intensive care unit population are recorded.

In an interim period an Alarm Advisor software will be introduced to the unit. In a second phase (post-implementation) the same set of alarm data will be recorded.

The "Alarm Advisor" Software can identify alarms based on criteria set by the medical staff and provide hints to reduce alarms and alarm nuisance (e.g. by proposing adjustments of alarm limits).

The effect of reduction of recurring nuisance alarms through the implementation of the Alarm Advisor shall be evaluated.

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted to the intensive care units during the study periods

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Routinely monitored intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 1336 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2018-03-11 (Actual)

PRIMARY OUTCOMES:
Number of Alarms | 2 month per phase with 2 month washout (6 month overall)
  red and yellow alarms with subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Funk, PhD, Professor, Principal Investigator — Yale School of Nursing
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No